CLINICAL TRIAL: NCT03057899
Title: Efficacy and Safety of a Mixed Extract of Fenugreek Seed and Lespedeza Cuneata in the Treatment of Testosterone Deficiency Syndrome: A Randomized, Double-blind, Placebo-Controlled Clinical Trial
Brief Title: Efficacy of Fenugreek Seed and Lespedeza Cuneata in TDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Jun Park, Associate Professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fenugreek for TDS
Record Dates: First submitted 2017-02-11; First posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Hypogonadism
Keywords: Herbal medicine; phytotherapy; testosterone
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fenugreek seed and Lespedeza cuneata (TFG) (Experimental): Patients who received investigational products (200 mg TFG) twice per day for 8 weeks at least 30 minutes after food intake
  Interventions: Drug: TFG capsules (200 mg /capsule)
- Placebo (Placebo Comparator): Patients who received placebo twice per day for 8 weeks at least 30 minutes after food intake
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: TFG capsules (200 mg /capsule) — TFG capsules were prepared using extracts from Trigonella foenum-graecum seed and Lespedeza cuneata. During the study period, two capsules were taken daily for 8 weeks.
  Other Names: mixed extract of fenugreek seed and Lespedeza cuneata (TFG)
  Arms: fenugreek seed and Lespedeza cuneata (TFG)
Drug: Placebo oral capsule — During the study period, two capsules were taken daily for 8 weeks. Placebo and TFG capsules were identical in shape, color, and taste.
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
Objective: The aim of this study was to investigate the efficacy and safety of a mixed extract of fenugreek seed and Lespedeza cuneata (TFG) for the treatment of testosterone deficiency syndrome (TDS).

Design: Patients were instructed to take a placebo capsule or 200 mg TFG capsule twice per day for 8 weeks.

Outcome measures: The primary efficacy variable was the change from baseline in the Aging Males' Symptoms scale (AMS), as well as levels of serum total testosterone and free testosterone. Secondary efficacy measurements included changes from baseline in the number of 'yes' answers on the Androgen Deficiency in the Aging Male questionnaire (ADAM), levels of serum total cholesterol, HDL-C, LDL-C, triglyceride, perceived stress scale (PSS-10), all domain scores of the International Index of Erectile Function (IIEF), as well as changes in body composition.

DETAILED DESCRIPTION:
Testosterone deficiency syndrome (TDS) is "a clinical and biochemical syndrome associated with advancing age and characterized by symptoms of a deficiency in serum testosterone levels". TDS can cause a significant decrease in quality of life and has many adverse effects on multiple organs in terms of men's health. In addition to the detrimental effect of sexual functions, men with TDS tend to have increased waist circumference, hyperglycemia, hypertriglyceridemia, hyperlipidemia, and a history of diabetes. TDS can be treated with testosterone replacement therapy (TRT). TRT should be initiated on an individualized basis in TDS patients who have clinical signs and symptoms of androgen deficiency if the benefits of treatment appear to outweigh the potential risks and only after thorough discussion with the patient. Different preparations of testosterone are currently available. The majority of clinical data shows that TRT is very safe and effective. There is currently no evidence that testosterone treatment increases the risk of prostate disease using modern guidelines. However, the fear of prostate cancer and the risk of erythrocytosis may represent the main limitations of TRT in aging men. Additionally, TRT cannot improve the function of Leydig cells (which produce testosterone), but only compensate for the lack of testosterone.

Limited research has focused on the use of herbal medicine to improve male health, particularly to increase testosterone levels and support healthy sexual function. Despite the increasing availability of effective conventional medical treatments, plant-derived and herbo-mineral remedies continue to be a popular alternative for men seeking to improve sexual function.

Trigonella foenum-graecum Linn, also known as fenugreek, is an aromatic annual plant that reaches heights of 30-60 cm. It is found wild in Kashmir, Punjab, and the upper Gangetic plains, and is widely cultivated in many parts of India. It is used internally as an abortifacient, antispasmodic, appetite stimulant, blood cleanser, laxative, tonic, and expectorant. It is also indicated externally for abscesses, boils, galactagogue, and for its demulcent and emollient properties. The seeds contain diosgenin along with three minor steroidal saponins (similagenin, savsalpogenin, and yuccagenin), choline, trimethylamine (a sex hormone in frogs), vitamins (A, B2, B6, B12, D), lysine, l-tryptophan rich proteins, mucilaginous fiber, coumarin, fenugreekine, nicotinic acid, sapogenins, phytic acid, scopletin and trigonelline, calcium, iron, β-carotene, and other vitamins and essential oils.

Previous studies have suggested that Trigonella foenum-graecum seed extract has positive effects on sexual health and quality of life, and that it demonstrates anabolic and androgenic activity in young patients. It is believed that these positive effects are due to increased testosterone, including free testosterone, and that Trigonella foenum-graecum seed extract may be an effective treatment for the symptoms of possible testosterone deficiency in aging men. The basis for this androgenic activity may be due to the fact that Trigonella foenum-graecum seeds contain soluble steroidal saponins, specifically furostanol glycosides, which are responsible for complexing cholesterol in the cell membrane. Other studies have found that Trigonella foenum-graecum increases testosterone and free testosterone, suggesting that it may be an incomplete 5-alpha reductase and aromatase inhibitor. The investigators investigated the efficacy and safety of a mixed extract of Trigonella foenum-graecum seed and lespedeza cuneata (TFG) for the treatment of TDS.

ELIGIBILITY:
Inclusion Criteria:

* total scores on the Aging Males' Symptoms scale (AMS) questionnaire ≥ 27; total serum cholesterol <220 mg/dl; and triglyceride 150-399 mg/dl

Exclusion Criteria:

* diagnosis of another sexual disorder, serum creatinine > 2.5 mg/dL, an uncontrolled psychiatric disorder, history of major hematological, renal, or hepatic abnormalities, body mass index ≥ 45 kg/m2, HBsAg (hepatitis B surface antigen) positive, prostate specific antigen (PSA) ≥ 4.0 ng/ml, cardiac failure, or a history of alcoholism or substance abuse. Patients who had taken PDE5 inhibitors, TRT, anti-androgen, statins, fibrates, niacin, steroid, fish oil, colestin, fiber-based laxatives, phytosterol margarines, anti-diabetics, anti-platelet, thyroxine, diuretics, or beta-blockers were also excluded.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Aging Males' Symptoms (AMS) scale | 4 week
level of serum total testosterone | 4 week
level of serum free testosterone | 4 week
Aging Males' Symptoms (AMS) scale | 8 week
level of serum total testosterone | 8 week
level of serum free testosterone | 8week

SECONDARY OUTCOMES:
percentage of positivity on the Androgen Deficiency in Aging Males (ADAM) questionnaire | 8 week
level of serum total cholesterol | 8 week
level of serum HDL-C | 8 week
level of serum LDL-C | 8 week
level of serum triglyceride | 8 week
perceived stress scale (PSS)-10 | 8 week
Scores of the International Index of Erectile Function (IIEF) | 8 week

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided